CLINICAL TRIAL: NCT05331677
Title: Correction of Multiplanar Deformities Around the Knee With Monolateral External Fixator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, mohamed mahmoud eldeeb, resident doctor at othopedic surgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-03-07
Record Dates: First submitted 2022-03-18; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Deformities Around the Knee in Pedietrics
MeSH Terms: interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental)
  Interventions: Procedure: correction of deformities around the knee with external fixator

INTERVENTIONS:
Procedure: correction of deformities around the knee with external fixator — minimally invasive surgery

SUMMARY:
Angular deformities around the knee are one of the common cause of presentation at pediatric orthopedic clinic. Although these conditions are commonly benign and self-limiting.

The mechanical axis of the lower extremity is a straight line extending from the center of the femoral head to the center of the ankle. The horizontal distance in millimeters from the center of the knee joint to the mechanical axis is the deviation of the mechanical axis.

The goal of treatment is to correct malalignment of the lower extremity and perhaps to prevent or delay the onset of osteoarthritis by normalizing the mechanical axis

ELIGIBILITY:
Inclusion Criteria:

* Genu valgus having tibio-femoral angle more than 15 degrees.
* Genu varus having metaphyseal-diaphyseal angle of more than 11 degrees
* More than one plane defirmity
* Age 10 - 16 yrs
* Range of motion:

  1. Full extension
  2. More than 100 in flextion

Exclusion Criteria:

* Genu recurvatum.
* Flexion deformity.
* Pathological conditions (e.g: bone softening diseases
* Dysplasia
* Limb length discrepancy

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Thoresen scoring system | one year
  * Malaligment varus/valgus procurvatum/retrocurvatum internal/external rotation
  * Range of motion flextion extension deficit pain and swelling

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Espandar R, Mortazavi SM, Baghdadi T. Angular deformities of the lower limb in children. Asian J Sports Med. 2010 Mar;1(1):46-53. doi: 10.5812/asjsm.34871. PMID 22375192
- [Background] Edgerton BC, Mariani EM, Morrey BF. Distal femoral varus osteotomy for painful genu valgum. A five-to-11-year follow-up study. Clin Orthop Relat Res. 1993 Mar;(288):263-9. PMID 8458142